CLINICAL TRIAL: NCT06163742
Title: A Phase I/II Randomized Trial to Determine the Safety of a Novel Donor Site Dressing (Product X)
Brief Title: Novel Donor Site Dressing (Product X)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16307
Record Dates: First submitted 2023-08-18; First posted 2023-12-11 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-02

CONDITIONS: Burns
Keywords: Donor Site; Burns; Wound Healing
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard-of-Care (Active Comparator)
  Interventions: Device: Standard-of-Care
- Product X (Experimental)
  Interventions: Device: Product X

INTERVENTIONS:
Device: Product X — The investigational device is a polyethylene glycol-based biomaterial. It can be applied to donor sites on the arms, torso, and legs.
  Arms: Product X
Device: Standard-of-Care — The active comparator includes the current standard-of-care treatment: hydrocellular polyurethane dressing covered with TegadermTM film for 48 hours, followed by an occlusive gauze impregnated with 3% Bismuth Tribromorphenate in petrolatum.
  Arms: Standard-of-Care

SUMMARY:
The goal of this clinical trial is to test a novel donor site dressing called Product X in burn patients requiring skin grafting procedures. A donor site is an area where the surgeon has taken a layer of skin to create a graft. This is required to make severe burn wounds heal. However, donor sites often experience infection, pain, and itch that can delay the healing of the donor site. To prevent these complications, donor sites are covered with dressings to prevent infection and absorb fluids from the wounds. Many options exist, but no single dressing is best, especially for pain management and the ability to absorb fluids from wounds effectively.

The investigators have developed a new donor site dressing to meet the criteria of an "ideal dressing," called Product X. The main question this clinical trial aims to determine the safety and potential wound-healing benefits of this donor site dressing as a new therapy that will help patients who require donor sites.

Participants will:

* Be randomized, like a flip of a coin, to receive either Product X or the standard-of-care dressings. If patients have one donor site, it will be randomized to receive either Product X or the standard-of-care dressings, Allevyn and Xeroform. If they have two donor sites, one donor site will be randomized to receive Product X and the other to receive standard-of-care dressings.
* Have photographs of their donor sites taken at the operation, during dressing changes, at discharge, and at regularly scheduled outpatient follow-up appointments with the burn clinic.
* Complete short questionnaires to assess their comfort (pain and itch) with their donor sites daily.
* Complete a scar formation questionnaire at your regularly scheduled follow-up appointments in the outpatient burn clinic.

Researchers will compare Product X to standard-of-care dressings (Allevyn and Xeroform) to see if there are improvements in wound healing, pain, itch, and infection.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age;
2. <25% total body surface area (TBSA) burn;
3. Deep partial or full-thickness burn requiring operative procedures;
4. Autologous donor site(s) on thigh, torso, and/or arm.

Exclusion Criteria:

1. Patients who are moribund.
2. Pregnancy.
3. Active cancer and currently undergoing treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of donor site infections | From date of donor site dressing application until date of hospital discharge, assessed up to 52 weeks.
  Donor site infection requiring antibiotic/antifungal treatment or additional (unplanned) OR.
Number of non-healing donor sites | From date of donor site dressing application until date of hospital discharge, assessed up to 52 weeks.
  Non-healing donor site requiring additional (unplanned) OR.
Poor scarring requiring additional (unplanned) OR measured with the Patient Observer Scar Assessment Score (POSAS). | At 3 months and 6 months post-hospital discharge.
  Scores will range from 1 to 10 for each measure, with higher scores indicating worse scarring.

SECONDARY OUTCOMES:
The amount of excess bleeding from the donor site measured by the need for interventions to control the bleeding. | From date of donor site dressing application until last dressing takedown, assessed up to 52 weeks.
Time from autografting procedure to 95% healing of donor site. | From date of donor site dressing application until hospital discharge, assessed up to 52 weeks.
  Photography and evaluation of the donor site at operation, dressing-take downs, and discharge from the hospital.
Scar formation over time using the Patient and Observer Scar Assessment Scale | At 3 months and 6 months post-hospital discharge.
  Scores will range from 1 to 10 for each measure, with higher scores indicating worse scarring.
Absorption of wound exudate measured daily by the amount of dressing required and the number of additional dressing changes needed. | From application of the donor site dressing until last dressing takedown, assessed up to 52 weeks.
  Greater amounts of dressings required and greater numbers of dressing changes indicate worse absorbability.
Number of patients experiencing adhesion of the dressing to the donor site | From application of the donor site dressing until last dressing takedown, assessed up to 52 weeks.
  Adhesion of the dressing to the donor site will be measured as: no adhesion, partial adhesion, or adhesion of the dressing to the donor site, with adhesion of the dressing to the donor site area having worse outcomes.
Range of motion of the donor site measured by the ability to actively participate in therapy sessions. | From application of the donor site dressing until last dressing takedown, assessed up to 52 weeks.
  Assessed in terms of the patient's subjective limitations in moving the donor site area. Measured as either: no limitations, minimal limitations, moderate limitations, or severe limitations in movement, with severe limitations being the worst outcome, indicating very limited movement of the donor site area.
Donor Site Pain | From application of the donor site dressing until last dressing takedown, assessed up to 52 weeks.
  Subjective donor site pain will be evaluated within 24 hours of each dressing change by participants using the Numeric Pain Scale. The Numeric Pain Scale ranges from 0 (no pain) to 10 (severe pain).
Itch | From application of the donor site dressing until last dressing takedown, assessed up to 52 weeks.
  Subjective measures of the presence and severity of itch will be measured daily by patients using the ItchyQuant scale, a validated numeric itch scale. The scale ranges from 0 (no itch) to 10 (severe itch).

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Jeschke, MD PhD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada